CLINICAL TRIAL: NCT00357500
Title: Anti-Angiogenic Chemotherapy: A Phase II Trial of the Oral 5-Drug Regimen (Thalidomide, Celecoxib, Fenofibrate, Etoposide and Cyclophosphamide) in Patients With Relapsed or Progressive Cancer
Brief Title: Etoposide, Cyclophosphamide, Thalidomide, Celecoxib, and Fenofibrate in Relapsed or Progressive Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Mark W. Kieran, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-343; P30CA006516 (NIH); CDR0000487628 (Other: NCI); NCT00165321 (obsolete NCT alias)
Record Dates: First submitted 2006-07-26; First posted 2006-07-27 (Estimated); Results first posted 2014-09-09 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Central Nervous System Tumor, Pediatric; Leukemia; Lymphoma; Neuroblastoma; Sarcoma; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: Metronomic; antiangiogenic
MeSH Terms: conditions — Central Nervous System Neoplasms; Leukemia; Lymphoma; Neuroblastoma; Sarcoma | interventions — Celecoxib; Cyclophosphamide; Etoposide; Fenofibrate; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 5-drug metronomic antiangiogenic regimen (Experimental): Thalidomide: Start at 3 mg/kg (rounded to nearest 50 mg), increasing dose weekly by 50 mg as tolerated to 24 mg/kg (max 1,000 mg); Celecoxib: < 20 kg at 100 mg; 20-50 kg at 200 mg; > 50 kg at 400 mg; Fenofibrate: 90 mg/m2 (max 200 mg); Etoposide: 50 mg/m2; Cyclophosphamide: 2.5 mg/kg (max 100 mg); Patients receive oral etoposide once daily on days 1-21 and 43-63 (weeks 1-3 and 7-9) and oral cyclophosphamide once daily on days 22-42 (weeks 4-6). Patients also receive oral thalidomide once daily, oral celecoxib twice daily, and oral fenofibrate once daily in weeks 1-9. Treatment repeats approximately every 9 weeks for at least 3 courses in the absence of disease progression or unacceptable toxicity. Patients receive alternating etoposide and cyclophosphamide pulses (i.e., etoposide-cyclophosphamide-etoposide during courses 1 and 3 and cyclophosphamide-etoposide-cyclophosphamide during course 2).
  Interventions: Drug: celecoxib; Drug: cyclophosphamide; Drug: etoposide; Drug: fenofibrate; Drug: thalidomide

INTERVENTIONS:
Drug: celecoxib
Drug: cyclophosphamide
Drug: etoposide
Drug: fenofibrate
Drug: thalidomide

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as etoposide and cyclophosphamide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Thalidomide, celecoxib, and fenofibrate may stop the growth of cancer cells by blocking blood flow to the cancer. Celecoxib also may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving combination chemotherapy together with thalidomide, celecoxib, and fenofibrate may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving etoposide and cyclophosphamide together with thalidomide, celecoxib, and fenofibrate works in treating young patients with relapsed or progressive cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the activity of etoposide, cyclophosphamide, thalidomide, celecoxib, and fenofibrate, in terms of prolonging the time to disease progression, in young patients with relapsed or progressive cancer.

Secondary

* Determine, preliminarily, the biologic activity of this regimen, in terms of tumor response and overall survival, in these patients.
* Determine the toxicity of this regimen in these patients.
* Evaluate different radiographic techniques as markers of tumor response in these patients.
* Evaluate the predictive ability of in vitro correlative studies as markers of tumor response.

STATISTICAL DESIGN: Patients were classified into one of 8 strata according to diagnosis: leukemia/lymphoma, bone tumors, neuroblastoma, high grade glial tumors, low grade glial tumors, ependymoma, medulloblastoma/PNET, and miscellaneous. A two-stage design for each disease stratum was planned. The accrual goal at the end of the two-stage design was 20 subjects for each stratum. A stopping rule was applied after the accrual of the first 10 eligible subjects enrolled in each disease stratum. If 1 or more patients in the first 10 evaluable patients were alive and progression-free at 27 weeks and have tolerated therapy then accrual to stage two would proceed. Among 20 patients within a stratum, if 3 or more patients met primary endpoint then regimen would be considered successful. The probability of concluding the treatment is feasible is 0.95 if true success rate is 30% and 0.07 if true succes rate is 5%. Overall accrual target was 80-160 patients. Please see published manuscript (Robison et al Pediatr Blood Cancer 2014) for results within disease strata.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed cancer (at diagnosis or relapse), including any of the following:

  * Leukemia and/or lymphoma (closed to accrual)
  * Bone tumor (e.g., Ewing's sarcoma or osteosarcoma) (closed to accrual)
  * Neuroblastoma (closed to accrual)
  * High-grade glial tumor
  * Low-grade glial tumor
  * Ependymoma
  * Medulloblastoma and/or primitive neuroectodermal tumor (PNET)
  * Miscellaneous tumor (closed to accrual)
  * Brain stem glioma, defined as intrinsic tumors of the pons causing diffuse enlargement

    * Brain stem glioma that progressed after radiotherapy does not require histological confirmation
    * Duration of symptoms at the time of diagnosis must be < 3 months

      * Symptoms should consist of cranial nerve deficits, ataxia, and/or long tract signs
* Relapsed or progressive poor prognosis disease for which no available curative therapy exists

PATIENT CHARACTERISTICS:

* Karnofsky performance status 50-100% OR Lansky play scale 50-100% (for infants)
* Life expectancy > 2 months
* Platelet count > 75,000/mm^3 (transfusion independent)
* Absolute neutrophil count > 1,000/mm^3 (in patients without bone marrow disease)
* Hemoglobin ≥ 9.0 g/dL
* Creatinine < 1.5 mg/dL OR creatinine clearance or glomerular filtration rate ≥ 70 mL/min
* Bilirubin ≤ 1.5 mg/dL
* SGPT ≤ 3 times normal
* SGOT ≤ 3 times normal (4 times normal for patients on ranitidine hydrochloride)
* Alkaline phosphatase ≤ 3 times normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double-method contraception during and for 2 months after completion of study treatment
* Must be willing to participate in the Celgene STEPS® program
* Recent thromboembolic disease (e.g., deep vein thrombosis or pulmonary embolism) allowed if patient is clinically stable and the thromboembolic event occurred > 3 weeks prior to study entry
* No active infection
* No active uncontrolled cardiac, hepatic, renal, or psychiatric disease ≥ grade 3
* No known allergies to sulfonamides
* No concurrent illness that would obscure toxicity or dangerously alter drug metabolism
* No other serious medical illness

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior therapy
* Prior chemotherapy and/or radiotherapy allowed
* Prior celecoxib allowed
* Prior standard-dose IV etoposide and cyclophosphamide administered in 3-week courses allowed
* No prior oral therapy with etoposide, thalidomide, cyclophosphamide, or fenofibrate for > 2 months in duration
* No other concurrent investigational agents
* No other concurrent nonsteroidal anti-inflammatory drugs
* Concurrent steroids and/or antiseizure medications allowed

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 101 (Actual)
Dates: Start 2005-01; Primary Completion 2013-02 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark W. Kieran, MD, PhD, Study Chair — Dana-Farber Cancer Institute
Locations (10):
- United States (10):
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Miami Children's Hospital, Miami, Florida
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Maine Medical Center Research Institute, Scarborough, Maine
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - St. Louis Children's Hospital, St Louis, Missouri
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - Hasbro Children's Hospital, Providence, Rhode Island

REFERENCES:
- [Background] Robison NJ, Campigotto F, Chi SN, Manley PE, Turner CD, Zimmerman MA, Chordas CA, Werger AM, Allen JC, Goldman S, Rubin JB, Isakoff MS, Pan WJ, Khatib ZA, Comito MA, Bendel AE, Pietrantonio JB, Kondrat L, Hubbs SM, Neuberg DS, Kieran MW. A phase II trial of a multi-agent oral antiangiogenic (metronomic) regimen in children with recurrent or progressive cancer. Pediatr Blood Cancer. 2014 Apr;61(4):636-42. doi: 10.1002/pbc.24794. Epub 2013 Oct 4. PMID 24123865

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was open for patient accrual at 11 different pediatric oncology centers from January 7, 2005 through March 6, 2009.
Pre-assignment Details: Patients must have recovered or stabalized the toxicity from prior therapy.
Period: Overall Study
Arm/Group | 5-drug Metronomic Antiangiogenic Regimen
Started | 101
Began Protocol Therapy | 97 (4 pts did not start treatment due either to removal of consent or inability to get insurance.)
Completed | 24
Not Completed | 77
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 5
Not completed — Progressive Disease | 65
Not completed — Not Started Protocol Therapy | 4

BASELINE CHARACTERISTICS:
Population: The analysis population represents patients who started treatment.
Groups:
- 5-drug Metronmic Antiangiogenic Regimen: Thalidomide: Start at 3 mg/kg (rounded to nearest 50 mg), increasing dose weekly by 50 mg as tolerated to 24 mg/kg (max 1,000 mg); Celecoxib: < 20 kg at 100 mg; 20-50 kg at 200 mg; > 50 kg at 400 mg; Fenofibrate: 90 mg/m2 (max 200 mg); Etoposide: 50 mg/m2; Cyclophosphamide: 2.5 mg/kg (max 100 mg); Patients receive oral etoposide once daily on days 1-21 and 43-63 (weeks 1-3 and 7-9) and oral cyclophosphamide once daily on days 22-42 (weeks 4-6). Patients also receive oral thalidomide once daily, oral celecoxib twice daily, and oral fenofibrate once daily in weeks 1-9. Treatment repeats approximately every 9 weeks for at least 3 courses in the absence of disease progression or unacceptable toxicity. Patients receive alternating etoposide and cyclophosphamide pulses (i.e., etoposide-cyclophosphamide-etoposide during courses 1 and 3 and cyclophosphamide-etoposide-cyclophosphamide during course 2).
Arm/Group | 5-drug Metronmic Antiangiogenic Regimen
Number analyzed (Participants) | 97
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 91
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 10 [0.52 to 21]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 50
Region of Enrollment [Number; unit: participants]
  United States | 97
Disease Group [Number; unit: participants] — Patients were stratified within 7 disease strata and an 8th 'miscellaneous' stratum.
  participants
    High Grade Glioma | 21
    Ependymoma | 19
    Low Grade Glioma | 12
    Bone Tumors | 12
    Medulloblastoma/PNET | 8
    Neuroblastoma | 3
    Leukemia/Lymphoma | 4
    Miscellaneous CNS Tumors | 9
    Miscellaneous non-CNS Tumors | 9

OUTCOME MEASURES:

1. Primary Outcome: Therapy Completion Rate
Description: Proportion of patients alive at 27 weeks without progressive disease (PD) and having tolerated therapy. As appropriate for tumor type and location, gadolinium-enhanced MRI and other imaging modalites were used to assess response. Progressive disease was defined as >/=25% increase in product of diameters, development of new areas of disease, or disease-attributable clinical deterioration or death, progressive disease. For patients with leukemia PD was defined as >/=25% or >/=5,000 cells/mm3 increase in number of circulating cells, development of extramedullary disease, or other clinical evidence of progression.
Time Frame: 27 weeks
Population: The analysis dataset is comprised of all treated patients.
Measure: Number (90% Confidence Interval); unit: proportion of patients
Arm/Group | 5-drug Metronomic Antiangiogenic Regimen
Number analyzed (Participants) | 97
proportion of patients | .25 [.18 to .33]

2. Secondary Outcome: 27-Week Progression-Free Survival
Description: 27-week progression-free survival is the probability of patients remaining alive and progression-free at 27-weeks from study entry estimated using Kaplan-Meier methods. As appropriate for tumor type and location, gadolinium-enhanced MRI and other imaging modalites were used to assess response. Progressive disease was defined as >/=25% increase in product of diameters, development of new areas of disease, or disease-attributable clinical deterioration or death, progressive disease. For patients with leukemia PD was defined as >/=25% or >/=5,000 cells/mm3 increase in number of circulating cells, development of extramedullary disease, or other clinical evidence of progression.
Time Frame: Assessed every 9 weeks on treatment and annually until death or initiation of new therapy, up to 27 weeks.
Population: The analysis dataset is comprised of all treated patients.
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | 5-drug Metronomic Antiangiogenic Regimen
Number analyzed (Participants) | 97
Probability | 0.31 [0.21 to 0.42]

3. Secondary Outcome: 27-Week Overall Survival
Description: 27-week overall survival is the probability of patients remaining alive at 27-weeks from study entry estimated using with Kaplan-Meier methods.
Time Frame: Assessed every 9 weeks on treatment and annually until death or initiation of new therapy, up to 27 weeks.
Population: The analysis dataset is comprised of all treated patients.
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | 5-drug Metronomic Antiangiogenic Regimen
Number analyzed (Participants) | 97
Probability | 0.61 [0.49 to 0.71]

4. Secondary Outcome: Best Response
Description: As appropriate for tumor type and location, gadolinium-enhanced MRI and other imaging modalites were used to assess response. Best response was regarded as best response at any single assessment. Response was defined as follows: complete resolution of all demonstrable tumor, complete response (CR); >/=50% decrease in the product of the 2 maximum perpendicular diameters relative to the baseline evaluation, partial response (PR); <50% decrease and <25% increase in product of diameters, stable disease (SD); and >/=25% increase in product of diameters, development of new areas of disease, or disease-attributable clinical deterioration or death, progressive disease (PD). For patients with leukemia PD was defined as >/=25% or >/=5,000 cells/mm3 increase in number of circulating cells, development of extramedullary disease, or other clinical evidence of progression.
Time Frame: Assessed at study entry, every 9 weeks on treatment and at treatment discontinuation, up to 27 weeks.
Measure: Number; unit: participants
Arm/Group | 5-drug Metronomic Antiangiogenic Regimen
Number analyzed (Participants) | 97
participants
  Complete Response | 1
  Partial Response | 12
  Stable Disease | 36
  Progressive Disease | 47
  Not Evaluable | 1

ADVERSE EVENTS:
Time Frame: 27 weeks
Arm/Group | 5-drug Metronomic Antiangiogenic Regimen
Serious Adverse Events (participants affected / at risk) | 74/97
Other Adverse Events (participants affected / at risk) | 81/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 5-drug Metronomic Antiangiogenic Regimen (N=97)
DE140 (General disorders) | 1
Death - disease progression NOS (General disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 21
Hematologic-other (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 9
Hearing w/w-o audiogr in monitor prg (Ear and labyrinth disorders) | 1
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 2
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 2
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Abdomen, pain (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 11
Fever w/o neutropenia (General disorders) | 1
Edema limb (General disorders) | 1
Extremity-lower (gait/walking) (General disorders) | 1
Infection w/ gr3-4 neut, catheter relate (Infections and infestations) | 1
Infection w/ gr3-4 neut, lung (Infections and infestations) | 2
Infection w/ gr3-4 neut, skin (Infections and infestations) | 1
Infection Gr0-2 neut, mucosa (Infections and infestations) | 1
Infection w/ unk ANC lung (Infections and infestations) | 1
Infection w/ unk ANC mucosa (Infections and infestations) | 1
Infection-other (Infections and infestations) | 1
Leukocytes (Investigations) | 57
Lymphopenia (Investigations) | 37
Neutrophils (Investigations) | 46
Platelets (Investigations) | 8
Alkaline phosphatase (Investigations) | 1
ALT, SGPT (Investigations) | 5
AST, SGOT (Investigations) | 3
Metabolic/Laboratory-other (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 1
Back, pain (Musculoskeletal and connective tissue disorders) | 1
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 1
Myelodysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ataxia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Neuropathy-motor (Nervous system disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 1
Psychosis (Psychiatric disorders) | 1
(ARDS) (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 5-drug Metronomic Antiangiogenic Regimen (N=97)
Myelodysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hemoglobin (Blood and lymphatic system disorders) | 52
Palpitations (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Cushingnoid appearance (Endocrine disorders) | 1
Neuropathy CN II vision (Eye disorders) | 1
Cataract (Eye disorders) | 1
Keratitis (Eye disorders) | 1
Ocular-other (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 16
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 8
Distention/bloating, abdominal (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 2
Hemorrhoids (Gastrointestinal disorders) | 1
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 3
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 20
Vomiting (Gastrointestinal disorders) | 12
GI-other (Gastrointestinal disorders) | 5
Anus, hemorrhage (Gastrointestinal disorders) | 1
Abdomen, pain (Gastrointestinal disorders) | 11
Anus, pain (Gastrointestinal disorders) | 1
Oral cavity, pain (Gastrointestinal disorders) | 1
Stomach, pain (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 31
Fever w/o neutropenia (General disorders) | 6
Rigors/chills (General disorders) | 2
Constitutional, other (General disorders) | 4
Edema limb (General disorders) | 1
Extremity-lower (gait/walking) (General disorders) | 1
Irritability (children <3yrs of age) (General disorders) | 1
Chest/thoracic pain NOS (General disorders) | 2
Pain-other (General disorders) | 3
Gallbladder, pain (Hepatobiliary disorders) | 1
Allergic reaction (Immune system disorders) | 1
Infection w/ gr3-4 neut, upper airway (Infections and infestations) | 3
Infection Gr0-2 neut, lip/perioral (Infections and infestations) | 1
Infection Gr0-2 neut, mucosa (Infections and infestations) | 1
Infection Gr0-2 neut, oral cavity (Infections and infestations) | 1
Infection Gr0-2 neut, upper airway (Infections and infestations) | 1
Infection w/ unk ANC oral cavity/gums (Infections and infestations) | 1
Infection Gr 0-2 neut, blood (Infections and infestations) | 1
Infection-other (Infections and infestations) | 3
Bruising (Injury, poisoning and procedural complications) | 1
Chemoradiation dermatitis (Injury, poisoning and procedural complications) | 1
Leukocytes (Investigations) | 18
Lymphopenia (Investigations) | 6
Neutrophils (Investigations) | 19
Platelets (Investigations) | 27
Weight gain (Investigations) | 2
Weight loss (Investigations) | 3
PTT (Investigations) | 1
Alkaline phosphatase (Investigations) | 7
ALT, SGPT (Investigations) | 32
AST, SGOT (Investigations) | 25
Bilirubin (Investigations) | 7
Creatinine (Investigations) | 5
Metabolic/Laboratory-other (Investigations) | 2
Obesity (Metabolism and nutrition disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 7
Dehydration (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 9
Bicarbonate (Metabolism and nutrition disorders) | 16
Hypercalcemia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 12
Hyperglycemia (Metabolism and nutrition disorders) | 18
Hypoglycemia (Metabolism and nutrition disorders) | 7
Hypermagnesemia (Metabolism and nutrition disorders) | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 7
Hyperkalemia (Metabolism and nutrition disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 5
Hypernatremia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 8
Musculoskeletal/soft tissue-other (Musculoskeletal and connective tissue disorders) | 1
Back, pain (Musculoskeletal and connective tissue disorders) | 1
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 4
Muscle, pain (Musculoskeletal and connective tissue disorders) | 1
Ataxia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 8
Memory impairment (Nervous system disorders) | 1
Neuropathy CN V jaw / face-sensory (Nervous system disorders) | 2
Neuropathy CN XII tongue (Nervous system disorders) | 1
Neuropathy-motor (Nervous system disorders) | 5
Neuropathy-sensory (Nervous system disorders) | 10
Pyramidal tract dysfunction (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 3
Speech impairment (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 2
Neurologic-other (Nervous system disorders) | 5
Head/headache (Nervous system disorders) | 7
Insomnia (Psychiatric disorders) | 1
Confusion (Psychiatric disorders) | 4
Agitation (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 3
Euphoria (Psychiatric disorders) | 1
Personality (Psychiatric disorders) | 4
Urinary hemorrhage NOS (Renal and urinary disorders) | 1
Hemoglobinuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Cystitis (Renal and urinary disorders) | 1
Incontinence urinary (Renal and urinary disorders) | 1
Renal/GU-other (Renal and urinary disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Muco/stomatitis by exam, pharynx (Respiratory, thoracic and mediastinal disorders) | 1
Muco/stomatitis (symptom) pharynx (Respiratory, thoracic and mediastinal disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 3
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 5
Dry skin (Skin and subcutaneous tissue disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 16
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 4
Rash/desquamation (Skin and subcutaneous tissue disorders) | 9
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Skin-other (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 3
Hypotension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less